CLINICAL TRIAL: NCT04637308
Title: A Randomized, Phase II Study of Succinylated Gelatin for Prevention of Fluid Retention in Patients With Breast Cancer Receiving Docetaxel Chemotherapy
Brief Title: Succinylated Gelatin for Prevention of Fluid Retention in Patients With Breast Cancer Receiving Docetaxel Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20190812
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Fluid Retention
Keywords: Fluid Retention; Chemotherapy; Succinylated gelatin; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — succinylated gelatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Succinylated gelatin (Experimental): The patients received intravenous infusion of succinylated gelatin one day before and on the day of chemotherapy, 500ml each time, once per day.
  Interventions: Drug: Succinylated gelatin
- Control (No Intervention): Observation.

INTERVENTIONS:
Drug: Succinylated gelatin — Succinylated gelatin (SG, "Gelofusine"; B. Braun, Crissier, Switzerland) is a clear, inexpensive, safe, colloidal plasma volume-expanding solution, weight-average molecular weight (MWw) 30 kDa.
  Arms: Succinylated gelatin

SUMMARY:
Breast cancer patients who received docetaxel chemotherapy were randomly divided into two groups; experimental group: the patients received intravenous infusion of succinylated gelatin one day before and on the day of chemotherapy, 500ml each time, once per day; control group: observation. Primary endpoint: total incidence of fluid retention. Secondary endpoints: severity and duration of fluid retention, change in quality of life score.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 years
* Diagnosed with breast cancer
* ECOG 0-2
* Received chemotherapy with docetaxel

Exclusion Criteria:

* Existed peripheral edema, ascites and pleural or pericardial effusion
* Serum creatinine exceeds 1.5 times of the upper normal limit
* Total serum bilirubin exceeds 1.25 times of the upper normal limit, or ASAT exceeds 2 times of the upper normal limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Total incidence of fluid retention | 6 months
  Total incidence of peripheral edema, ascites and pleural or pericardial effusion of patients during the period of docetaxel chemotherapy

SECONDARY OUTCOMES:
severity of fluid retention | 6 months
  Severity of peripheral edema, ascites and pleural or pericardial effusion of patients during the period of docetaxel chemotherapy; the severity of pain was evaluated by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, ranging from 1 to 3 grades.
change in Functional Assessment of Cancer Therapy-Breast subscale score | 6 months
  Functional Assessment of Cancer Therapy-Breast（FACT-B）subscale during the period of docetaxel chemotherapy was assessed; the scores range from 0 to 144, higher scores mean a better outcome (higher quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China